CLINICAL TRIAL: NCT06532617
Title: A Single-arm Phase II Clinical Study of Cadonilimab Combined With S-1 or Capecitabine as Second-line Treatment for Patients With Advanced Pancreatic Cancer
Brief Title: Cadonilimab Combined With S-1 or Capecitabine as Second-line Treatment for Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang Long, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240515024702669
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Neoplasms
Keywords: PD-1/CTLA-4 Bispecific Antibody
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+S-1or Capecitabine (Experimental)
  Interventions: Drug: Cadonilimab+S-1or Capecitabine

INTERVENTIONS:
Drug: Cadonilimab+S-1or Capecitabine — Eligible patients will receive Cadonilimab (6mg/k, iv, D1,Q3W)combined with S-1 (40-60mg po BID Q3W D1-14）or Capecitabine (1250mg/m2, po BID Q3W D1-14）until disease progression or unacceptable toxicity. Patients who had used S-1 in the first line should choose capecitabine; patients who had used capecitabine in the first line should choose S-1; otherwise decided by investigator's choice.

SUMMARY:
This is a single arm, single cencer, phase II clinical trial. This study aims to evaluate the efficacy and safety of Cadonilimab combined with S-1 or capecitabine as a second-line treatment for advanced pancreatic cancer.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed written informed consent
* Age 18-80, female or male
* Histopathologically confirmed pancreatic ductal adenocarcinoma
* Patients with locally advanced pancreatic cancer who have previously received standard first-line anti-tumor treatment (radiotherapy, chemotherapy, targeted or immunotherapy, etc.)
* Locally advanced pancreatic cancer is defined as follows: a. The tumor has no distant metastasis; b. Pancreatic head/uncinate process: The tumor contacts the superior mesenteric artery >180˚; c. Pancreatic body and tail: The tumor contacts the superior mesenteric artery or celiac artery >180˚; The tumor contacts the celiac artery and infiltrates the abdominal aorta; d. The tumor invades the jejunal branch of the superior mesenteric artery. Portal vein-superior mesenteric vein cannot be safely reconstructed due to tumor invasion, vein occlusion, or involvement of a large range of jejunal branches of the superior mesenteric vein.
* At least one measurable lesion (RECIST1.1)
* ECOG PS 0-1
* Expected survival time>3 months
* Adequate organ function

Main Exclusion Criteria:

* Malignant diseases other than pancreatic cancer diagnosed within 5 years before the first dose (excluding radically resected basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ)
* Currently participating in interventional clinical research treatment, or having received other research drugs or used research devices within 4 weeks before the first dose
* Active autoimmune disease
* Allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Allergic to the active ingredients or excipients of this study drug, cadonilimab, S-1 or capecitabine
* Have not fully recovered from any toxicity and/or complications caused by the intervention before starting treatment
* History of HIV
* Active HBV or HCV
* Pregnant or breastfeeding women
* Any severe or uncontrolled systemic disease
* Active pulmonary tuberculosis
* People with mental disorders who are unable to cooperate with treatment
* Uncontrolled infection
* The investigators assess that the subjects are unable to complete the entire trial process or are otherwise unsuitable for participating in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Defined as the proportion of patients with a complete response or partial response to treatment according to RECIST1.1

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  Defined as the length of time from the first dose to death from any cause.
Progression-free survival (PFS) | Up to 2 years
  Defined as the length of time from the first dose to progression disease or death from any cause.
Disease control rate (DCR) | Up to 2 years
  Defined as the proportion of patients with a complete response, partial response or stable disease to treatment according to RECIST1.1
Duration of response (DoR) | Up to 2 years
  Defined as the length of time from first tumor response (CR or PR) to disease progression (PD) or death.

OTHER OUTCOMES:
Biomarker analysis | Up to 2 years
  Biomarkers that potentially predict efficacy include, but are not limited to, PD-L1 expression and T cell subpopulations in tumor tissue specimens or blood samples and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China